CLINICAL TRIAL: NCT02935751
Title: Apixaban Discontinuation Prior to Major Surgery
Acronym: ADIOS
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: 16G.421
Record Dates: First submitted 2016-10-14; First posted 2016-10-17 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Hemorrhage; Thromboembolism
MeSH Terms: conditions — Hemorrhage; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Lab tests for plasma levels of apixaban and anti-10a factor — All patients will have a blood draw at 48 hours prior to elective surgical procedure and then a second blood draw on the morning of the procedure to test apixaban plasma and anti-Xa levels.

SUMMARY:
The ADIOS study is a prospective, observational study will evaluate one hundred and thirty (130) patients with non-valvular atrial fibrillation who are currently receiving treatment with apixaban as indicated to reduce the risk of stroke or systemic embolism, and who require an elective major surgical or invasive procedure will be included in the study. The purpose of the study is to evaluate the efficacy of the recommended pre-procedure washout period of 48 hours.

DETAILED DESCRIPTION:
This study will estimate for what proportion of patients a 48 hour pre-procedure apixaban discontinuation is sufficient to achieve minimal apixaban plasma levels (less than 30 ng/mL) prior to surgery. The investigators hypothesize that this portion will be 80-95%.

All patients will have a blood draw at 48 hours prior to procedure and then a second blood draw on the morning of the procedure to test apixaban plasma and anti-Xa levels. Patients will also receive a follow-up phone call at 30 days to collect information on clinical events.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* On long term anticoagulation with apixaban for treatment of non-valvular atrial fibrillation or venous thromboembolism
* Undergoing elective major surgery or invasive procedure

Exclusion Criteria:

* Inability to obtain informed consent for the blood sample draws
* Any condition precluding collection of follow-up information
* Participation in another clinical trial
* Apixaban Package Insert Recommendations and Cautions
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.
* Women must not be breastfeeding
* WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug apixaban plus 5 half-lives of study drug apixaban (approximately 3 days) plus 30 days (duration of ovulatory cycle) for a total of 33 days post- treatment completion.
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug apixaban plus 5 half-lives of the study drug (approximately 3 days) plus 90 days (duration of sperm turnover) for a total of 93 days post-treatment completion.
* Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However WOCBP must still undergo pregnancy testing as described.
* The safety and efficacy of apixaban have not been studied in patients with prosthetic heart valves. Therefore, use is not recommended in these patients.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 130 patients who are currently receiving treatment with apixaban for non-valvular atrial fibrillation and scheduled for an elective surgical procedure.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-07 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Apixaban plasma concentration | Prior to elective surgery
  Determine whether the recommended 48 hour pre-procedure discontinuation period is sufficient to achieve minimal apixaban plasma concentration of < 30 ng/ml prior to surgery

SECONDARY OUTCOMES:
Anti-10a apixaban plasma concentration | Prior to elective surgery
  Assess changes in anti-Xa apixaban levels following apixaban discontinuation but prior to the procedure
30 day outcomes assessment | Up to 30 days post- procedure
  Incidence of major events within 30 days including bleeding events, arterial thromboembolic events, and deaths caused by bleeding or thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Geno J. Merli, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Merli GJ, Kraft WK, Eraso LH, Galanis T, Thomson LJ, Ouma GO, Viscusi E, Gong JZ, Lam E. Apixaban Discontinuation for Invasive Or major Surgical procedures (ADIOS): A prospective cohort study. Vasc Med. 2022 Jun;27(3):269-276. doi: 10.1177/1358863X211047270. Epub 2021 Nov 22. PMID 34809507